CLINICAL TRIAL: NCT03553719
Title: Enhancing European Management of Analgesia, Sedation and Delirium - Implementation and Validity of Pain, Agitation and Delirium Screening in the ICU - an International, Prospective Multicenter Observational Trial
Brief Title: Enhancing European Management of Analgesia, Sedation and Delirium
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: EuMAS
Record Dates: First submitted 2018-04-24; First posted 2018-06-12 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- One day point-prevalence analysis 1: Data on the management of intensive care unit patients ≥18 years will be collected. Data of approximately 170 patients per point-prevalence analysis will be collected.
- One day point-prevalence analysis 2: Before the start of the second one day point-prevalence analysis a training package is conducted at each study center. This contains online lectures, instructional videos, educational handouts, and a bedside teaching component over the course of 6 weeks. The effect of a training block for intensive care unit staff on routine delirium screening rate and the change of the other outcome measures will be assessed.
  During the one day point-prevalence analysis 2 data on the management of intensive care unit patients ≥18 years will be collected. Data of approximately 170 patients per point-prevalence analysis will be collected.
- One day point-prevalence analysis 3: Data on the management of intensive care unit patients ≥18 years will be collected. Data of approximately 170 patients per point-prevalence analysis will be collected.

SUMMARY:
This prospective, multicenter study aims to evaluate the effect of routine training of intensive care unit (ICU) staff on the implementation rate of screening tools for pain, agitation and delirium (PAD) ) in three one day point-prevalence analyses.

The evaluations will take the form of one day point-prevalence analyses, administered both pre- and post-training phase.

The 6-week training block consists of e-learning material in the form of text content, slides and brief training videos.

At each point-prevalence analysis, data of approximately 300 patients in 14 participating centers will be collected.

Data collection focuses primarily on parameters of routine patient management (e.g. medications, screening scores) and basic patient characteristics (e.g. illness severity, age, major comorbidities).

Additionally, one member of each major profession in the ICU care team (attending physician, resident physician, nurse) will be given a brief online questionnaire to gauge their estimate of routine practice with regards to delirium screening and delirium prevalence in their ICU.

Each participating patient will also receive one "gold standard" delirium screening with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU score) performed by a trained expert.

DETAILED DESCRIPTION:
ICU-staff that is adequately trained in PAD-screening and -management is part of guideline recommendations internationally, and staff training should take place accordingly. Prior studies have hinted at low implementation rates of delirium screening intensive care units and an overall low reliability of the documented scores.

The study's rationale is to evaluate staff perceptions regarding delirium screening practice in their ICU, and evaluate the validity of routine delirium screening scoring (compared to an expert-screen). Subsequently, the effect of a training block for ICU staff on routine delirium screening frequency and validity will be assessed.

The implemented training package contains online lectures, instructional videos, educational handouts, and a bedside teaching component over the course of 6 weeks.

On each point-prevalence day three members of the ICU staff (attending/consultant, trainee physician, nurse) will fill out their respective questionnaire (attending CRF, physician CRF, nurse CRF). These questionnaires ask for estimates of delirium prevalence in their respective ICU, as well as estimates on the frequency of delirium screening implementation.

Subsequently, the local study coordinator will evaluate all patients that have received treatment in the ICU during the past 24 hours according to the inclusion and exclusion criteria. Each included patient will receive a pseudonym and the study coordinator will fill out one electronic case report file (eCRF, see list of items) per included patient.

A member of staff who is trained in administering the CAM-ICU screening tool will then evaluate all included patients, and enter the respective score result in each patient's "expert CRF".

ELIGIBILITY:
Inclusion criteria:

* Patient treated in the intensive care unit
* Age ≥18 years

Exclusion criteria:

* Blindness
* Deafness
* Lack of relevant language skills to complete assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data on the management of ICU patients ≥18 years will be collected. Data of approximately 170 patients per point-prevalence analysis will be collected. As the main parameters in question concern the routine patient management, there will be no follow-up on individuals
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Delirium screening rate | Up to 24 hours
  The delirium screening rate is documented and calculated according to patients´ records.

SECONDARY OUTCOMES:
Delirium screening rate | Up to 24 hours
  The rate of occurrence of delirium screening of some form is documented according to the estimation by clinical staff: One member of each major profession in the ICU care team (attending physician, trainee physician, nurse) will be given a brief online questionnaire to gauge their estimate of routine practice with regards to delirium screening and delirium prevalence in their ICU.
Delirium screening type - as documented in the patient chart | Up to 24 hours
  During each point prevalence analysis, one investigator at each study site will search the respective patient charts for documentation of delirium screening type used and the scores during the preceding 24 hours.
Delirium screening score - as documented in the patient chart | Up to 24 hours
  During each point prevalence analysis, one investigator at each study site will search the respective patient charts for documentation of delirium screening scores during the preceding 24 hours.
Confusion assessment method for the intensive care unit (CAM-ICU) | Up to 24 hours
  CAM-ICU form patient records
Confusion assessment method for the intensive care unit (CAM-ICU) scoring by trained expert | Up to 24 hours
  Each participating patient will receive one "gold standard" delirium screening with the CAM-ICU score performed by a trained expert. Each participating patient will receive one "gold standard" delirium screening with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score performed by a trained expert.
  The test assesses a patient's state of confusion and serves as a screening test for ICU-related delirium.
  The tested patient can either be "positive" or "negative" for delirium, or "not testable", if the patient's state of consciousness does not allow administration of the test.
Extracorporeal organ support | Up to 24 hours
  The type of extracorporeal organ support measures that a patient received on the day of analysis, as well as during the course of his ICU stay before the day of analysis will be documented.
Parameters of infection | Up to 24 hours
  The patient's sepsis status according to SIRS- as well as Sepsis-3-criteria on the day of analysis will be documented.
Use of relevant medication | Up to 24 hours
  The use of sedatives, analgesics, antipsychotics, vasopressors and inotropes during the day of analysis will be documented, as well as their daily cumulative dose.
Daily cumulative dose of relevant medication | Up to 24 hours
  The daily cumulative dose of sedatives, analgesics, antipsychotics, vasopressors and inotropes during the day of analysis will be documented,
Mobilization | Up to 24 hours
  The type of mobilization measures that a patient received on the day of analysis will be documented, ranging from passive in-bed mobilization, to active mobilization in-bed or sitting, to ambulation.
Relevant non-pharmacologic measures | Up to 24 hours
  The occurrence of non-pharmacologic measures to treat and/or prevent delirium during the patient's ICU stay will be documented. Options include: noise-reduction, light therapy, and also a free-text option to add other modalities.
Family involvement | Up to 24 hours
  Occurrence of caregiver and/or family talks during the patient's ICU stay will be documented.
Sedation score | Up to 24 hours
  The type of sedation screening and the patient's score on the day of analysis will be documented. The Richmond Agitation Sedation Scale measures a patient's state of sedation on a scale from -5 (not arousable) to +4 (agitated, combative), with 0 implying an awake and calm patient.
Pain assessment type on day of analysis | Up to 24 hours
  The type of pain assessment tool and the patient's score on the day of analysis will be documented.
  Different centers might used different tools to assess patient's pain level. This item asks each center to name the scoring tool used for the patient.
Pain screening score on day of analysis | Up to 24 hours
  The the patient's pain screening score on the day of analysis will be documented.
  The achievable score depends on the screening instrument used in the participating centers.

OTHER OUTCOMES:
Acute Physiology And Chronic Health Evaluation (APACHE II) - Score | At the beginning of the investigation
  The Acute Physiology And Chronic Health Evaluation (APACHE II) score is a classification system for disease severity for ICU patients. The score is calculated using 12 measurements from routine ICU patient management, as well as the patient's age. The scores range from 0-71, with higher scores corresponding to higher disease severity and mortality risk.
Sequential Organ Failure Assessment (SOFA) - Score | At the beginning of the investigation
  The Sequential Organ Failure Assessment score (SOFA) is a tool commonly used in the ICU to assess the patient's risk for morbidity and mortality. It contains 6 values from routine ICU management, each being scored on a scale from 0-4.
  Thus, a patient can have SOFA scores ranging from 0 to 24, with higher scores corresponding to higher risk.
Age | At the beginning of the investigation
Gender | At the beginning of the investigation
Height | At the beginning of the investigation
Weight | At the beginning of the investigation
Major comorbidities | At the beginning of the investigation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Univ. - Prof. Dr. med. Claudia Spies, Mitte, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paul N, Grunow JJ, Rosenthal M, Spies CD, Page VJ, Hanison J, Patel B, Rosenberg A, von Haken R, Pietsch U, Schrag C, Waydhas C, Schellongowski P, Lobmeyr E, Sander M, Piper SK, Conway D, Totzeck A, Weiss B. Enhancing European Management of Analgesia, Sedation, and Delirium: A Multinational, Prospective, Interventional Before-After Trial. Neurocrit Care. 2024 Jun;40(3):898-908. doi: 10.1007/s12028-023-01837-8. Epub 2023 Sep 11. PMID 37697129